CLINICAL TRIAL: NCT05104593
Title: An Integrated Solution for Sustainable Care for Multimorbid Elderly Patients With Mild Cognitive Impairment or Mild Dementia (CAREPATH)
Brief Title: An Integrated Solution for Sustainable Care for Multimorbid Elderly Patients With Dementia
Acronym: CAREPATH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Collaborators: ECLEXYS SAGL (Unknown); The Fraunhofer-Gesellschaft (Other); Klinikum Bielefeld (Other); University of Warwick (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); University of Castilla-La Mancha (Other); CENTRUL IT PENTRU STIINTA SI TEHNOLOGIE (Unknown); SRDC YAZILIM ARASTIRMA VE GELISTIRME VE DANISMANLIK TICARET ANONIM SIRKETI (Unknown); OCTILIUM SAGL (Unknown)
Responsible Party: Principal Investigator, Pedro Abizanda, Principal Investigator, Complejo Hospitalario Universitario de Albacete
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAREPATH; 945169 (Other Grant/Funding Number: European Commission, H2020-SC1-2020-Two-Stage-RTD)
Record Dates: First submitted 2021-10-21; First posted 2021-11-03 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Comorbidities and Coexisting Conditions; Alzheimer Disease; Dementia; Malnutrition; Frailty; Sarcopenia; Stroke; Asthma; Chronic Obstructive Pulmonary Disease; Chronic Kidney Diseases; Heart Failure; Diabetes; Coronary Artery Disease; Hypertension; Behavioral Symptoms
Keywords: Alzheimer Disease; Dementia; Quality of Life; Multimorbidity; Health monitoring; Home monitoring; Telemedicine
MeSH Terms: conditions — Alzheimer Disease; Dementia; Malnutrition; Frailty; Sarcopenia; Stroke; Asthma; Pulmonary Disease, Chronic Obstructive; Renal Insufficiency, Chronic; Heart Failure; Diabetes Mellitus; Coronary Artery Disease; Hypertension; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: Randomization will be performed centrally using a computerized system that uses stratified block randomization. After screening, patients who meet all eligibility criteria will be randomly assigned to 1 of 2 treatment groups (CAREPATH or control). Patients will be randomized in a CAREPATH to control ratio of 1:1. Randomization to intervention allocation will be stratified by sex, associated comorbidity and geographic region. Stratification factors will ensure balance of these factors across intervention arms and facilitate unbiased estimate of intervention effect in subgroups.
Who Masked: Outcomes Assessor
Masking Description: The study is to be conducted in a simple-blind manner to minimize potential bias from investigators. It is not possible to conduct a double-blind study, because patients will know if they are using CAREPATH or not. In each site, two different investigators will be involved in the study. The first one will be responsible of initial assessments, randomization and management during follow-up. The investigator responsible of follow-up assessments for outcomes will be blinded to the assignment group in order to reduce the treatment effect bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention tested (CAREPATH) (Experimental): The intervention tested will be the CAREPATH system.
  Interventions: Other: Intervention tested (CAREPATH)
- Control group (No Intervention): Control group, no intervention

INTERVENTIONS:
Other: Intervention tested (CAREPATH) — The intervention tested will be the CAREPATH system. CAREPATH consists of an integrated, patient-centred, flexible and modular system that will provide a viable solution for the improvement of the management of multimorbid elderly patients with Mild Cognitive Impairment or mild dementia, with the help of clinicians. CAREPATH will act on patients and their informal caregivers, and its main objective is to empower multimorbid patients with MCI or mild dementia to manage their health condition together with their informal caregiver by providing assistance and reinforcement to follow their individual care plans, so independence and quality of life will increase for both of them. The intervention will provide a personalized care plan and activities proposal (treatment, activities proposal, lifestyle changes, referrals etc.) to patients and caregivers, considering the various sources of patient data available through the CAREPATH platform, and with the help of clinicians.
  Arms: Intervention tested (CAREPATH)

SUMMARY:
The CAREPATH will conduct Technical Validation and Usability (TVU) study by involving ≥ 45 target end users (16 patients with MCI or mild dementia with their informal caregivers and 16 healthcare professionals from various disciplines) and Clinical Investigation (CI) study involving ≥ 200 patients (≥ 100 users to pilot the CAREPATH platform and ≥ 100 patients as reference cases). Both of these pilot studies will be coordinated in four European countries (Spain, Romania, Germany and UK) with diverse health and social care systems, ICT landscape/digital maturity of healthcare provision and dementia national programs, which will allow for strengthening the evidence base on health outcomes and efficiency gains.

The CAREPATH outcomes can be summarized as:

1. An Integrated Care Platform that jointly addresses multimorbidity, dementia and diminished intrinsic capacity and optimally manages healthcare interventions for its users (patients, informal caregiver, healthcare providers, etc).
2. Technical Validation and Usability (TVU) study involving over 45 users and Clinical Investigation (CI) involving over 200 patients that will be conducted in four European countries (Spain, Romania, Germany and UK) during two years and mobilizing the other necessary actors, such as caregivers and healthcare professionals, for the validation of healthcare interventions.
3. Dementia / Multimorbidity Guidelines that will be conceived for best healthcare delivery.
4. Health Economics Impact Assessment for healthcare cost effectiveness and care provision equalities. The incremental cost-effectiveness and the incremental cost-utility ratio would allow revealing the incremental cost (or the potential savings) per unit of benefit of switching from usual care to CAREPATH-an integrated patient-centred approach- in multimorbid elderly patients with dementia, and therefore, to determinate whether the CAREPATH approach would be considered as a cost-effective alternative.

DETAILED DESCRIPTION:
The study will have two parts:

A. Usability study In order to ensure that the CAREPATH system is well-usable by its main target user groups namely patients with Mild Cognitive Impairment (MCI) or mild dementia, their informal caregivers and health care professionals in charge of caring for this patient group, a usability evaluation of the platform will be conducted as part of the Technical Validation and Usability (TVU) study described in chapter 1.3.6 of the proposal (IEC TR 62366-2: 2016-04 Medical devices - Part 2: Guidance on the application of usability engineering to medical devices). It will be carried out at the end of the main development phase to investigate usability issues and its results will serve as input for the (re-)design of the platform before the clinical investigation starts. Implementation of good usability of a medical device such as the CAREPATH platform is also enforced by the usability engineering process required now in the development of a medical devices by the new Medical Device Regulation (Regulation (EU) 2017/745) (Regulation (EU) 2017/745 of the European parliament and of the council of 5 April 2017 on medical devices, amending Directive 2001/83/EC, Regulation (EC) No 178/2002 and Regulation (EC) No 1223/2009 and repealing Council Directives 90/385/EEC and 93/42/EEC) which originates in the concern that increasing complexity and interactivity of medical devices bears a high risk of errors in handling if poorly designed causing harm to patients. Therefore, usability and safety are seen as interrelated and in the CAREPATH usability study possible hazardous situations will also be taken into account.

B. Clinical Investigation with a Medical Device class IIa After finishing the TVU, a Clinical Investigation will be conducted in order to validate the technological system CAREPATH for multimorbid elderly patients with MCI up to mild dementia (see Work Package 5 of the complete proposal). This version of CAREPATH will include the modifications made by engineers in the system after the analysis of the TVU phase.

The main objective will be to analyze the reduction in healthcare appointments and the hypothesis is that CAREPATH will improve Quality of Life (QoL) of these patients through a multicomponent approach based on the 5 following principles:

1. Identification of purpose.
2. Establishment of disease and treatment burden, by considering how a person's health problems affect their day-to-day life, their mental health and their wellbeing.
3. Formulation of patient goals, values and priorities
4. Communicating to patients and caregivers the benefits, risks and costs of treatments and medications.
5. Provision of an individualised care plan.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged ≥ 65 years old (randomization will warrant that at least 40% of each sex will be included in the study).
* Meets NIAAA core clinical criteria for probable Alzheimer disease, dementia or Mild Cognitive Impairment due to Alzheimer´s Disease (consistent with the NIAAA diagnostic criteria and guidelines for MCI; Albert MS, DeKosky ST, Dickson B, et al. The diagnosis of mild cognitive impairment due to Alzheimer's disease: Recommendations from the National Institute on Aging Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimer's & Dement 2011; 7: 270-9)
* Mild symptomatology, as defined by a screening MMSE score of ≥ 22 points and CDR-GS of 0.5 or 1.0.
* Evidence of retrospective decline in cognitive functions.
* Multimorbidity: Presence of at least one of the following chronic diseases: Diabetes mellitus needing pharmacologic treatment, hypertension needing pharmacologic treatment, heart failure NYHA class 2-4, atrial fibrillation with a CHA2DS2-Vasc, chronic obstructive pulmonary disease (COPD) GOLD staging B-D, asthma needing pharmacologic treatment or chronic kidney disease (CKD) stage III-V.
* Living at home.
* Independence for basic activities of daily living.
* Availability of a person (referred to as the "caregiver" throughout this protocol) who in the investigator's judgment:

  * Has frequent and sufficient contact with the patient to be able to provide accurate information regarding the patient's cognitive and functional abilities, agrees to provide information at clinic visits (which require partner input for scale completion), signs the necessary consent form, and has sufficient cognitive capacity to accurately report upon the patient's behavior and cognitive and functional abilities.
  * Is in sufficiently good general health to have a high likelihood of maintaining the same level of interaction with the patient and participation in study procedures throughout the study duration.
  * Note that every effort should be made to have same caregiver participate throughout the duration of the study.
* Fluency in the language used at the study site.
* Willingness and ability to complete all aspects of the study; the patient should be capable of completing assessments either alone or with the help of the caregiver.
* Adequate visual and auditory acuity, in the investigator's judgement, sufficient to perform the neuropsychological testing (eye glasses and hearing aids are permitted).
* Patient must have completed at least 6 years of formal education after the age of 5 years.
* Able to provide written consent signed by the patient (co-signed by the patient's legally authorized representative, if required by the local regulations, guidelines, and independent ethics committee or institutional review board [IRB]).

  * Patients should be judged by the investigator to be lucid and oriented to person, place, time, and situation when giving the informed consent.
  * In judging capacity, the investigator must confirm that the patient is able to understand the information relevant to the decision to participate in the study, appreciate the situation in terms of the treatment and research options and their likely outcomes, and weigh the potential risks and benefits of participation in order to come to a decision and communicate that decision.

Exclusion Criteria:

* Any evidence of established dementia, including but not limited to, frontotemporal dementia, dementia with Lewy bodies, vascular dementia, Parkinson's disease, corticobasal degeneration, Creutzfeldt-Jakob disease, progressive supranuclear palsy, frontotemporal degeneration, Huntington's disease, normal pressure hydrocephalus, seizure disorder, or hypoxia. Presence of cerebral tumors, trauma, infections, autoimmune diseases or vitamin deficits (B12, folate…) affecting cognition.
* At risk of suicide in the opinion of the investigator.
* Inadequate home infrastructure to host the required technology.
* Inability to understand how to use the CAREPATH system.
* Illness that impedes carrying out the study:

  * Active cancer of any type except non-melanoma skin cancer.
  * Terminal disease (<12 months of life expectancy).
  * Other pathologies involving clinical instability.
* Psychiatric disorders or alcohol/drugs abuse.
* Living with a participant.
* Participation in other interventional clinical studies

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in healthcare appointments | 1 year
  The following healthcare appointments will be recorded, including if they are scheduled or unscheduled, date, reason, actions taken and relationship with CAREPATH.
  Hospitalization Emergency visits Outpatient specialists visits at hospital or in polyclinics Primary care/General Practitioners medical visit Primary care nurse visit At-home medical visit At-home nurse visit Physiotherapist or occupational therapist visit Psychologist/Psychiatry visit Nutritionist/Dietist visit Radiology tests Lab analysis Other clinical tests

SECONDARY OUTCOMES:
Quality of Life (QoL) | 1 year
  QoL will be determined using the EuroQoL-5D test, validated for these populations (Balestroni G, Bertolotti G. EuroQol-5D (EQ-5D): an instrument for measuring quality of life.
Change in unplanned care | 1 year
  Reduction in unplanned care: Unplanned care will be considered when the appointment to the service is not programmed at least 48 hours in anticipation, except for institutionalization or day centre admission.
Change in inappropriate prescription | 1 year
  Decrease in inappropriate prescription: STOPP/START criteria will be used to assess inappropriate prescription medicines (O´Mahony D, O´Sullivan D, Byrne S, et al. STOPP/START criteria for potentially inappropriate prescribing in older people: versión 2; Age Ageing 2015; 44: 213-18).
Change in number of participants with advanced directives | 1 year
  Increased number of participants with advanced directives: Written document available for advanced decisions for healthcare. The document should be agreed upon patient, Primary Care Physician/ General Practitioner and main caregiver to be considered valid for outcomes assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request. Study protocol, statistical analysis and clinical study report will be shared when data will be published in a Journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At data Journal publication